CLINICAL TRIAL: NCT03444168
Title: Central Nervous System Amplification in Lumbar Failed Back Surgery Syndrome
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: STUDY00140263; 1K23GM123320-01 (NIH)
Record Dates: First submitted 2018-02-08; First posted 2018-02-23 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
Keywords: lumbar spine surgery; lumbar failed back surgery syndrome
MeSH Terms: conditions — Chronic Pain; Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Candidate for Lumbar Spine Surgery: Participants have been designated to be a candidate for lumbar spine surgery to treat chronic low back and/or leg pain and you have agreed to proceed with the surgery.
- Lumbar Failed Back Surgery Syndrome: Participants have been diagnosed with having lumbar failed back surgery syndrome and have persistent and moderate-to-severe low back and/or leg pain for more than 6 months after a lumbar spine surgery.
- Healthy Volunteer: Participants are a healthy volunteer wishing to participate in a research study.

SUMMARY:
The purpose of this study is to learn whether or not certain risk factors and patient characteristics are linked with and possibly can predict the development of chronic pain after lumbar spine surgery.

ELIGIBILITY:
Inclusion Criteria For All Participants:

* Ability to read and speak English to allow for written informed consent, phenotyping, and patient-reported outcomes measures

Exclusion Criteria For All Participants:

* Individuals receiving or applying for compensation or disability and other aspects associated with potential secondary gain
* Inability to provide written informed consent
* Severe physical impairment
* Co-morbid medical conditions that may significantly impair physical functional status
* Illicit drug or unreported opioid use
* Medical or psychiatric conditions that in the judgment of study personnel would preclude participation in this study
* Pregnant or nursing
* Liver failure
* Self-reported liver cirrhosis
* Self-reported hepatitis
* Severe Cardiovascular disease

Inclusion Criteria for Candidates for Lumbar Spine Surgery:

* Deemed to be a candidate for primary lumbar spine surgery including but not limited to: lumbar laminectomy, discectomy, and fusion/instrumentation
* Diagnostic clinical and radiographic findings including but not limited to: lumbar degenerative disc disease, lumbar disc protrusion, herniation, or extrusion, lumbar spondylosis, lumbar spinal stenosis, lumbar spondylolisthesis or spondylolysis
* Willingness to participate in longitudinal follow-up or 6-months after their surgery.

Exclusion Criteria for Candidates for Lumbar Spine Surgery:

* History of previous lumbar spine surgery
* Indication for lumbar spine surgery is due to spinal cancer-related diagnosis
* Need for urgent or emergent lumbar spine surgery

Inclusion Criteria for Candidates with Lumbar Failed Back Surgery Syndrome:

* Chronic low back pain (+/- leg pain) for >= to 6 months duration after lumbar spine surgery (with or without instrumented fusion)
* Low back pain severity is moderate to severe (Numerical Rating Scale [NRS] Score >=4)

Exclusion Criteria for Candidates with Lumbar Failed Back Surgery Syndrome:

* Have a structural spinal lesion that would make them a current candidate for a revision lumbar spine surgery

Inclusion Criteria for Healthy Volunteers:

* No major diseases or diagnoses influencing pain or function

Exclusion Criteria for Healthy Volunteers:

* No chronic pain condition
* Score 3 or greater on the 2011 FM Survey Criteria (i.e. individuals with very mild fatigue or sleep problems will be allowed to participate as this is extremely common in the general population)

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited directly by the Candidate and by referral from specialist physicians at the KUMC Marc A. Asher, MD, Comprehensive Spine and Pain Management Center.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Clinical pain severity | Change from Baseline to Month 6
  Measured by the Brief Pain Inventory (BPI). The BPI scores are a numerical rating scale and range from 0 to 10. A score of 0 is equal to no pain and a score of 10 is equal to pain as bad as you can imagine.

SECONDARY OUTCOMES:
PROMIS (Patient-Reported Outcomes Measurement Information System) | Change from Baseline to Month 6
  PROMIS measures to be included are Depression, Anxiety, Physical Functioning, Fatigue, Sleep Impairment, Emotional Support, and Social Participation. Each questionnaire usually has 4-16 response options ranging in value from one to five. The total raw score for a short form with all questions answered is the sum of the values of the response to each question. The total range of potential raw scores depends on the number of questions being asked, for example, a 6 item form would have a range from is 6 to 30. After the raw score is calculated, a T-score metric is used to convert the raw score to a T-score. On the T-score metric, a score of 50 is the mean of a relevant reference population and 10 is the standard deviation of that mean. For PROMIS measures, higher scores equals "more of the concept being measured", this could be a desirable or undesirable outcome, depending on the concept being measured.
Oswestry Disability Index | Change from Baseline to Month 6
  The Oswestry Disability Index will be used to assess low back pain. There are 10 sections on the index. Each section has a possible score of 5. The total possible range of scores is 0 to 50. A score of 0 indicates no pain. A score of 50 indicates the person is bed-bound or exaggerating their symptoms.
2011 Fibromyalgia Survey | Change from Baseline to Month 6
  A measure of symptom severity in fibromyalgia. There is a total range of scores from 0 to 31. The higher the score the more severe a person's symptoms.

OTHER OUTCOMES:
Magnetic Resonance Imaging - Brain Regions and Pain Processing | Baseline
  A subgroup of patients enrolled will also undergo four different neuroimaging procedures (all in one visit) to identify brain regions and associated neurotransmitters operative in pain processing and modulation.
Quantitative Sensory Testing (QST) - Pressure pain sensitivity by Algometry | Baseline
  Pressure pain sensitivity is measured by Algometry (measured at the trapezius and lumbar spine). It yields a pressure pain threshold value measured in kPA.
Quantitative Sensory Testing (QST) - Pressure pain sensitivity by Multimodal Automated Sensory Testing | Baseline
  Pressure pain sensitivity is measured by the Multimodal Automated Sensory Testing (MAST) System (measured at the thumbnail). It yields a pressure pain threshold value measured in kg/cm2.
Quantitative Sensory Testing (QST) - Cuff Algometry | Baseline
  Cuff Algometry as measured by a rapid cuff inflator (measured at the gastrocnemius muscle). It yields a deep pressure pain threshold as measured in mmHg.
Quantitative Sensory Testing (QST) - Conditioned Pain Modulation (CPM) | Change from Post-stimulus test at Baseline visit to Pre-stimulus test at Baseline visit
  Conditioned Pain Modulation as measured at the thumbnail using the MAST. It yields a numerical pain rating difference on a 0-100 numerical scale that can either be positive or negative called CPM magnitude. CPM magnitude will be calculated as the difference (post-pre) in the mean of the three pain ratings given to the test stimulus prior to the conditioning stimuli and the three pain ratings of the test stimulus given during the conditioning stimuli. A reduction in test stimulus rating by conditioning stimulation implies functional (inhibitory) CPM, and the degree of reduction expresses the efficiency of CPM.
Wind Up Ratio (WUR) | Baseline
  Temporal Summation as measured at the forearm and the lumbar spine using a PinPrick Algometer. It yields a numerical pain rating score from 0-100 numerical scale that will then be used to calculate the Wind Up Ratio (WUR) which is the mean pain rating of three stimulus trains divided by the mean pain rating of a single stimuli. A WUR >1 indicates temporal summation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Chadwick, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States